CLINICAL TRIAL: NCT04918979
Title: Triage Information Extraction Technology Development and Database Construction for Emergent Patients Based on Voice and Image Recognition Technology
Brief Title: Information Extraction and Database Construction for Emergent Patients Based on Voice and Image Recognition Technology
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Collaborators: National Research Foundation of Korea (Other)
Responsible Party: Sponsor
Other Study IDs: SNUEMSAVTR
Record Dates: First submitted 2021-06-01; First posted 2021-06-09 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-05

CONDITIONS: Emergencies
Keywords: Triage; Emergency department; Voice recognition; Image recognition
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Video and audio data of the triage process of emergency department (ED) patients will be collected to build a database. Clinical information retrieved from the database with voice and image technology will be used to determine the triage level of each patient and will be compared with the actual triage level.

DETAILED DESCRIPTION:
Study Objectives:

1. To develop a platform to record video and audio data of the ED triage process.
2. To retrieve clinical information using voice and image technology.
3. To develop a tool to determine ED triage level using voice and image technology.
4. To build a clinical database using video and audio data using voice and image technology.

Study design: Single center observational study (tertiary hospital emergency department in Korea).

A platform to record video and audio data of the ED triage process will be developed. The camera and microphone will be installed at an optimal location to retrieve video and audio data in the ED triage area.

Voice and image technology will be used to retrieve clinical information including demographic information, chief complaint, type and onset of symptoms, past medical history, and physical examination results to build a database. Clinical information including examination notes, diagnosis, patient vital signs, test results, and ED results will be retrieved from the hospital database.

ELIGIBILITY:
Inclusion Criteria:

* Age 19 years or older
* Visited the emergency department of the study hospital

Exclusion Criteria:

* Patients who do not agree to enroll to this study
* Without a family
* Foreign patients

Min Age: 19 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adults who visit the emergency department without one of the exclusion criteria will be enrolled in this study.
Sampling Method: Non-Probability Sample
Enrollment: 428 (Actual)
Dates: Start 2020-02-12 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
The degree of agreement between emergency department triage level retrieved using voice/image technology and by nurses/physicians. | At the time of study completion (May 2022 anticipated).
  Korean triage and acuity scale (KTAS) which was developed based on Canadian triage and acuity scale (CTAS) is used in Korea. KTAS is composed of 5 levels: level 1, resuscitation; level 2, emergent; level 3, urgent; level 4, less urgent; level 5, non-urgent. Emergency department triage level will be assessed by using voice/image technology and will be compared with the triage level assessed by nurses/physicians. The triage level will be assessed during emergency department triage.

CONTACTS AND LOCATIONS:
Overall Officials: Ki Jeong Hong, PhD, Study Director — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea